CLINICAL TRIAL: NCT06564896
Title: Comparing A Conventional CPAP Airsense 10 VS Portable Air-Mini CPAP For Obstructive Sleep Apnea From Users' Perspective; A Cross - Over Study
Brief Title: Conventional CPAP Airsense 10 VS Portable Air-Mini CPAP For Obstructive Sleep Apnea (CASPAM)
Acronym: CASPAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FF-2024-303
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CPAP Airsense 10 (Active Comparator): Participants in CPAP Airsense 10
  Interventions: Device: CPAP Airsense 10 vs Air-Mini
- CPAP AIr-Mini (Active Comparator): Participants in CPAP AIr-Mini
  Interventions: Device: CPAP Airsense 10 vs Air-Mini

INTERVENTIONS:
Device: CPAP Airsense 10 vs Air-Mini — Patients' satisfaction and CPAP efficacy

SUMMARY:
Obstructive sleep apnea (OSA) has been one of the topmost global health problems. It is an underdiagnosed disease which have a huge burden on healthcare if left untreated. Almost 80-90% of adults are underdiagnosed of OSA Obesity primarily is one of the supreme risk factors for developing OSA. Globally, obesity cases have risen affecting almost two billion people. According to National Health and Morbidity Survey (NHMS) 2019, 1 in 2 adults in Malaysia were overweight or obese. Report from World Obesity Atlas 2023 predicts that adult obesity will rise 4.7% annually from 2020 - 2035, while child obesity will increase by 5.3% per year over similar timeline. Overweight individuals will have a significant economic impact on Malaysia's Gross Domestic Product (GDP) by 2035 by 2.8% which is estimated to be about RM 3.2 trillion.

Sequalae of OSA is divided into two (cardiovascular-metabolic effect and neurocognitive effect). This group of patients are at high risk of developing hypertension, insulin resistance, dyslipidemia which then leads to pulmonary hypertension and heart failure. More importantly, from the neurocognitive point of view, persistent sleep deprivation will lead to poor concentration, impaired memory, personality changes affecting overall self-performance which can lead to depression and compromising safety as they have higher risk of work-related accidents.

DETAILED DESCRIPTION:
Hypothesis

1. Participants' overall satisfaction is better using Air-Mini CPAP compared to Airsense CPAP machine.
2. There is no difference in terms of AHI reduction and average 95th centile pressure required between AirMini CPAP compared to Airsense CPAP machine.
3. There will be positive correlation between overall satisfaction and AHI reduction for Air-Mini CPAP compared to Airsense CPAP machine.
4. There is improvement in air leak, comfort, compactness and maintenance in AirMini CPAP machine compared to AirSense CPAP.

This is a prospective cross over trial study of group of patients with moderate to severe OSA based on the severity of the AHI.

This study will be conducted for all moderate to severe OSA participants in Hospital Canselor Tuanku Muhriz (medical and non-medical department) between September 2024 to December 2026.

This is a cross over trial that includes patients with medium to high risk of OSA according to STOPBANG score. Once these group of participants are selected, consent will be taken from them to go through a scheduled sleep study. Diagnosis is established after AHI score is concluded from the polysomnographic study. Those who are diagnosed with moderate to high AHI score will be recruited in this study. All subjects will be given a CPAP trial using both AirSense and AirMini model for 7 days each device. Upon recruitment, the subject will be randomised using 1:1 block randomisation either to receive AIrsense 10 CPAP machine or Air-mini CPAP machine.

Those participants that use AirSense CPAP machine first for 7 days will be given a set of Questionnaire at the end of 7th day of the trial. Subsequently, they will be switch to use Air-Mini CPAP machine for another 7 days and the same set Questionnaire will be given on the 7th day of the trial. The type of the interface used will be based on subject's preferences, i.e., full face mask / nasal masak / nasal pillow, during the initial 1 - 2 days of CPAP trial. The same interface as per subject's preferences will be used throughout the CPAP trials for both AirSense as well as Airmini CPAP machine.

The Questionnaire given comprises of a 100mm Visual Analogue Score (VAS) for: 1) Overall satisfaction, 2) Air Leak, 3) Comfort, 4) Compactness & Portability, 5) Maintenance & Configuration.

The data collected will be analyzed using SPSS Version 27.

This is a cross-sectional prospective study; hence the sample size calculation will be based on Machin et al. (2018) The sample size decided for this study was 40 subjects. Considering and taking into account of about 10% dropout / missing data, hence the total sample size that will be recruited for this study are 50 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Patients diagnosed with moderate to severe OSA (based on AHI classification from sleep study performed).
* Patients who are able to understand and answer the questionnaire given.

Exclusion Criteria:

* Patients who are unable to give consent to the study.
* Patients who have been diagnosed with OSA and already on CPAP machine.
* Patients who had underlying Obesity Hypoventilation Syndrome (OHS).
* Patients who had underlying co-morbidities that worsen apnea symptoms, such as congestive cardiac failure, active malignancy, narcolepsy, active alcohol or drug abuse, treatment-refractory dementia, psychotic illness and active use of drugs that disturb the sleep architecture (i.e hypnotics or stimulants of central nervous system).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the overall satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving conventional CPAP Airsense 10 (0 mm - Not Satisfied at all, 100mm - Very Satisfied) | 7 days after first usage of CPAP Airsense 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsence 10
To compare the overall satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Air-Mini. (0 mm - Not Satisfied at all, 100mm - Very Satisfied) | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Air Mini

SECONDARY OUTCOMES:
To evaluate the efficacy of CPAP machine Airsense 10 in terms of percentage AHI reduction (Optimal titration=AHI <5, Good titration=AHI ≤10 or by 50%, Adequate titration= AHI reduction by 75% from baseline) | 7 days after first usage of CPAP Airsense 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsense 10
To evaluate the efficacy of CPAP machine Air-Mini 10 in terms of percentage AHI reduction (Optimal titration=AHI <5, Good titration=AHI ≤10 or by 50%, Adequate titration= AHI reduction by 75% from baseline) | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Air-Mini
To determine the average 95th centile pressure required using conventional CPAP Airsense 10 | 7 days after first usage of CPAP Airsence 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsence 10
To determine the average 95th centile pressure required using CPAP Air-Mini | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Air-Mini
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving conventional CPAP Airsense 10 (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of air leak | 7 days after first usage of CPAP Airsence 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsence 10
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Air Mini (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of air leak | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using Air-Mini
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Airsense 10 (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of comfort | 7 days after first usage of CPAP Airsence 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsence 10
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Air-Mini (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of comfort | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Air-Mini
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Airsense 10 (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of compactness & portability | 7 days after first usage of CPAP Airsence 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsence 10
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Air-Mini (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of compactness & portability | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Air-Mini
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Airsense 10 (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of maintenance & configuration | 7 days after first usage of CPAP Airsence 10
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Airsence 10
To compare the satisfaction using Visual Analogue Score 100mm among moderate to severe OSA participants receiving CPAP Air-Mini (0 mm - Not Satisfied at all, 100mm - Very Satisfied), in terms of maintenance & configuration | 7 days after first usage of CPAP Air-Mini
  Participants with moderate to severe OSA who underwent CPAP trial using CPAP Air-Mini

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, MBBS(IIUM), Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Faculty of Medicine, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbasi A, Gupta SS, Sabharwal N, Meghrajani V, Sharma S, Kamholz S, Kupfer Y. A comprehensive review of obstructive sleep apnea. Sleep Sci. 2021 Apr-Jun;14(2):142-154. doi: 10.5935/1984-0063.20200056. PMID 34381578
- [Result] Ryan S, Taylor CT, McNicholas WT. Systemic inflammation: a key factor in the pathogenesis of cardiovascular complications in obstructive sleep apnoea syndrome? Thorax. 2009 Jul;64(7):631-6. doi: 10.1136/thx.2008.105577. PMID 19561283
- [Result] Rotenberg BW, Vicini C, Pang EB, Pang KP. Reconsidering first-line treatment for obstructive sleep apnea: a systematic review of the literature. J Otolaryngol Head Neck Surg. 2016 Apr 6;45:23. doi: 10.1186/s40463-016-0136-4. PMID 27048606

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT06564896/Prot_ICF_000.pdf